CLINICAL TRIAL: NCT06260007
Title: Efficacy and Safety Study of Products Based on Tribulus Terrestris, L. in Men With Oligospermia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRIHER0323OR-IV
Record Dates: First submitted 2023-11-28; First posted 2024-02-14 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia | interventions — Tribulus extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tribulus terrestris 94mg (Experimental)
  Interventions: Drug: Tribulus terrestris
- Tribulus terrestris 280mg (Experimental)
  Interventions: Drug: Tribulus terrestris
- Tribulus terrestris 250mg (Experimental)
  Interventions: Drug: Tribulus terrestris
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tribulus terrestris — Tribulus terrestris
  Arms: Tribulus terrestris 250mg; Tribulus terrestris 280mg; Tribulus terrestris 94mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Efficacy and Safety of Products Based on Tribulus terrestris, L. in Men with Oligospermia. It is expected that the benefits of investigational products outweigh the risks that will be mitigated or carefully managed by the study team.

ELIGIBILITY:
Inclusion Criteria:

1. - Male;
2. - Ages 25 and 60;
3. - Diagnosis of oligospermia;
4. - With sexual partner;
5. - Indication of drug treatment with steroid hormones, precursors or analogues.

Exclusion Criteria:

1. - Severe oligospermia
2. - Anatomical change
3. - Previous treatment for oligospermia or concomitant treatment with steroid, anabolic, hormonal precursors such as testosterone or analogues;
4. - BMI 35;
5. - Participant who presents liver enzyme and creatinine values above the upper limit of normality;
6. - History of testicular cancer, or prostate cancer or any other condition that carries risks in this case increased testosterone;
7. - Hypersensitivity to any ingredient present in the formulation;
8. - Any criteria or clinical history that, in the investigator's opinion, could compromise the well-being and participant safety;
9. - Proven infertility of the partner;
10. - History of genetic disorder;
11. - History of psychiatric disorder, serious or decompensated illness or any situation that, Investigator's discretion, puts the participant's safety at risk;
12. - Active cancer at the discretion of the Investigator;
13. - Participants with pregnant and breastfeeding partners;
14. - Cycling and horse riding more than 3 hours per week;
15. - Alcoholism characterized by the inability to control alcohol consumption according to WHO "drinker excessive, whose dependence on alcohol is accompanied by mental, health and physics, relationships with others and social and economic behavior". Source: https://www.cancer.gov/publications/dictionaries/cancerterms/def/alcoholism;
16. - Smoking greater than half a pack per day or equivalent.

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08-17 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of each product in men with changes in their spermogram compared to placebo. | 3 months
  Any improvement in sperm concentration (n/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Brasil Pesquisa Científica E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No